CLINICAL TRIAL: NCT06410859
Title: A Randomized, Double-blind, Parallel, Placebo-controlled, Multicenter, Phase 2 Clinical Trial to Evaluate the Efficacy, Safety, and Immunogenicity of Botulinum Toxin Type A for Injection (HengLi®) in the Treatment of Trigeminal Neuralgia
Brief Title: Botulinum Toxin Type A for Injection (HengLi®) in the Treatment of Trigeminal Neuralgia
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: LKGS_277 (Industry)
Responsible Party: Sponsor-Investigator, LKGS_277, Linna Wang , director, Lanzhou Institute of Biological Products Co., Ltd
Organization: Lanzhou Institute of Biological Products Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HengLi009-Ⅱ
Record Dates: First submitted 2024-04-14; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Trigeminal Neuralgia
Keywords: Botulinum Toxin Type A for Injection (HengLi®)
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Botulinum Toxin Type A for Injection(5U/site） (Experimental): 5U/site
  Interventions: Drug: Botulinum Toxin Type A for Injection,also known as "HengLi®"
- Botulinum Toxin Type A for Injection（2.5U/site） (Experimental): 2.5U/site
  Interventions: Drug: Botulinum Toxin Type A for Injection,also known as "HengLi®"
- placebo (Experimental): 0U/site
  Interventions: Drug: Botulinum Toxin Type A for Injection,also known as "HengLi®"

INTERVENTIONS:
Drug: Botulinum Toxin Type A for Injection,also known as "HengLi®" — This study plans to enroll 240 subjects, and the efficacy measures [VAS score, DSIS score, daily pain duration (if applicable), and number of daily pain episodes] will be collected from subjects using the electronic Patient-Reported Outcomes (ePRO) throughout the study. The study period mainly consists of a screening period (14 days before the first dose), a double-blind treatment period (from the first dose to Week 12), and an extension period (from Week 13 to Week 52), including a maximum of 4 treatment cycles (each cycle lasts 12 week)

SUMMARY:
To evaluate the efficacy of different dosing regimens of Botulinum Toxin Type A for Injection (HengLi®) in the treatment of trigeminal neuralgia (TN), so as to determine the optimal dosing regimen of the best administration scheme of Botulinum Toxin Type A for Injection (HengLi®) in the treatment of TN.

DETAILED DESCRIPTION:
This study plans to enroll 240 subjects, and the efficacy measures [VAS score, DSIS score, daily pain duration (if applicable), and number of daily pain episodes] will be collected from subjects using the electronic Patient-Reported Outcomes (ePRO) throughout the study. The study period mainly consists of a screening period (14 days before the first dose), a double-blind treatment period (from the first dose to Week 12), and an extension period (from Week 13 to Week 52), including a maximum of 4 treatment cycles (each cycle lasts 12 week)

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign the written ICF;
2. Male or female 18 to 75 years of age (inclusive), able to provide legal identification;
3. Subjects clinically diagnosed as classical or idiopathic TN, with pain in one or two divisions (diagnostic criteria in the International Classification of Headache Disorders, 3rd Edition [ICHD-3], see Appendix 6);
4. Have a mean daily VAS score of ≥ 40 mm for 7 consecutive days during the screening period, with mean number of daily episodes ≥ 2, and duration of pain ≥ 3 months at screening;
5. Have a clear consciousness, the ability to perceive and resolve pain, the ability to understand and cooperate with the clinical study process, and the ability to comply with the requirements of the study protocol until completion of the study;
6. Prior first-line drug therapy (carbamazepine, oxcarbazepine) for TN;
7. Women of childbearing potential (WOCBP) should have a negative pregnancy test within 7 days prior to the first dose, and subjects and their partners should have no pregnancy plan and promise to use a medically acceptable contraceptive measure (e.g., intrauterine device [IUD], contraceptive pill or condom) during the study drug treatment period and within 3 months after the last dose of study drug; Note: WOCBP is defined as non-postmenopausal women who have experienced menarche and have not undergone sterilization (hysterectomy or bilateral adnexectomy) or other causes of permanent infertility (e.g., mullerian agenesis) identified by investigator. Postmenopause is defined as amenorrhea for ≥12 months without other biological or physiological causes.

Exclusion Criteria:

1. Subjects with TN who have a history of surgical treatment, such as percutaneous radiofrequency thermocoagulation of trigeminal ganglion, Meckel's cave compression, stereotactic gamma knife radiotherapy. and microvascular decompression;
2. Change in the dose and type of drugs for treatment of TN changed within 4 weeks prior to the first dose (including carbamazepine, oxcarbazepine, gabapentin, lamotrigine, etc.);
3. Subjects who have received injection therapy (magnesium sulfate injection), physical therapy, or traditional Chinese medicine treatment of TN within 4 weeks prior to the first dose, such as ultrashort wave, magnetic therapy, acupuncture, traditional Chinese medicines, etc.;
4. Patients who have received any botulinum agent within 6 months prior to the first dose;
5. Patients with secondary TN confirmed by magnetic resonance imaging (MRI);
6. Patients with systemic neuromuscular junction disorders, such as myasthenia, Eaton Lambert syndrome, amyotrophic (spinal cord) lateral sclerosis, multiple sclerosis, etc.;
7. Subjects who have used drugs affecting neuromuscular junction within 7 days prior to the first dose (for example, aminoglycoside antibiotics [e.g., gentamycin, etc.], quinine, and penicillamine) or need to use the above drugs, cholinesterase antagonists, succinylcholine, curare-like depolarizing antagonists, magnesium sulfate, quinidine, calcium channel blockers (excluding antihypertensive agents such as amlodipine besylate and nifedipine), lincomycin, polymyxin, etc. during the conduct of the clinical trial;
8. There are conditions that investigator believes may affect pain assessment, such as skin disorders in the affected skin areas and may affect sensation, or the recommended injection sites have localized infection or are locally accompanied by other skin disorders;
9. Concurrent or prior hemorrhagic conditions, or intake of anticoagulants [e.g. heparin, coumarins, non-vitamin K antagonists, oral anticoagulants (e.g., apixaban, dabigatran, edoxaban, rivaroxaban), but aspirin and other platelet aggregation inhibitors such as ticlopidine, clopidogrel, prasugrel, abciximab, eptifibatide, and tirofiban are allowed] within 10 days prior to injection;
10. Chronic systemic diseases, which may affect subject's participation in the study as assessed by investigator, including but not limited to:

1）、Severe cardiopulmonary diseases, such as unstable angina pectoris, myocardial infarction, and severe arrhythmia, World Health Organization (WHO) cardiac function classification of Class III to IV at screening, hypertension poorly controlled with active treatment, systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg at the time of screening; recurrent asthmatic attacks, etc.; 2）、Cerebrovascular accident (e.g., cerebral infarction, transient ischemic attack, etc.) within 6 months prior to screening; 3）、History of malignant tumor (excluding cured skin basal cell carcinoma, carcinoma in situ, and papillary thyroid carcinoma) or history of anti-tumor treatment within 5 years prior to screening; 4）、Other severe or unstable medical conditions (such as systemic infection, lung diseases, liver, cardiovascular, kidney or gastrointestinal diseases, etc.) assessed by investigator; 11、Severe hematological, liver, and renal dysfunction, with any one of the following clinical laboratory test results:

1. 、Hematology: neutrophil count (ANC) < 1.5 × 109/L, or platelet count < 90 × 109/L, or hemoglobin < 100 g/L;
2. 、Hepatic function: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 × upper limit of normal (ULN); or total bilirubin (TBIL)> 1.5 × ULN;
3. 、Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 (calculated according to the simplified MDRD formula); 12、Presence of nervous/mental system disorders, which, in the investigator's opinion, may affect the evaluation of TN or self-scoring, including psychiatric disorders such as epilepsy, recurrent dizziness, headache, memory and cognitive impairment, severe depression, and schizophrenia, or other nervous system disorders except TN, such as headache and migraine; 13、Pregnant women and subjects in pregnancy or lactation; 14、Patients with known hypersensitivity to botulinum toxin type A and any ingredient in the formulation (sucrose, dextran, and gelatin) or with an allergic constitution; 15、Use of prohibited medications (see Section 6.5. 2) prior to screening. If a subject has used any prohibited medication before screening, screening is not allowed unless medication have been discontinued for at least 5 half-lives (see the labeling for the specific half-life) before the signing of ICF, and the medication is prohibited throughout the study; 16、Known history of drug/alcohol abuse; 17、Hepatitis B virus deoxyribonucleic acid (HBV-DNA) higher than the upper limit of detection, hepatitis C virus antibody (HCV-Ab) and HCV ribonucleic acid (RNA) positive, human immunodeficiency virus antibody (HIV Ab) positive, and serum Treponema pallidum antibody (TPPA method) positive at screening, or any of them; 18、Corneal ulcer; 19、Other conditions that make use of botulinum therapy unsuitable or may damage the safety of subjects or may make it impossible to complete the study in compliance with the protocol, as assessed by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of different dosing regimens of Botulinum Toxin Type A for Injection (HengLi®) in the treatment of trigeminal neuralgia (TN), so as to determine the optimal dosing regimen of the best administration scheme of BoNTA | Week 12
  Change in mean visual analogue scale (VAS) score at Week 12 from the mean VAS score over one week at baseline.
  for VAS,Pain was scored on a scale of 0 to10, with 0 indicating no pain, 10 indicating severe pain, and the middle part indicating varying degrees of pain.

SECONDARY OUTCOMES:
To evaluate the duration of response to different dosing regimens of Botulinum Toxin Type A for Injection (HengLi®) in the treatment of TN. | week4,week 8
  Changes in the mean visual analogue scale (VAS) scores of Week 4 and 8 of the double-blind treatment period from the mean VAS score over one week at baseline;
To evaluate the duration of response to different dosing regimens of Botulinum Toxin Type A for Injection (HengLi®) in the treatment of TN. | week4,week 8,week 12
  Changes in the mean number of daily pain episodes at Week 4, 8, and 12 of the double-blind treatment period from the mean number of daily pain episodes over one week at baseline;
To evaluate the duration of response to different dosing regimens of Botulinum Toxin Type A for Injection (HengLi®) in the treatment of TN. | week4,week8,week 12
  Changes in mean daily pain duration of subjects with persistent pain over one week [only those with persistent pain (such as dull pain) judged by investigator] at Week 4, 8, and 12 of the double-blind treatment period from the mean daily pain duration over one week at baseline;
To evaluate the duration of response to different dosing regimens of Botulinum Toxin Type A for Injection (HengLi®) in the treatment of TN. | week4,week 12
  Effect of the investigational product versus placebo on Patient Global Impression of Change (PGIC, Appendix 2) at Week 4 and 12 of the double-blind treatment period;PGIC is a 7-point scale reporting the patient's overall improvement in pain status:(1)very much improved;(2)much improved;(3)minimally improved;(4)no change;(5) minimally worse;(6)much worse;(7)very much worse
To evaluate the duration of response to different dosing regimens of Botulinum Toxin Type A for Injection (HengLi®) in the treatment of TN. | week4,week8,week 12
  Proportions of subjects with ≥ 50% and ≥ 30% reductions in mean visual analogue scale (VAS) score at Week 4, 8, and 12 of the double-blind treatment period from the mean VAS score over one week at baseline;for VAS,Pain was scored on a scale of 0 to10, with 0 indicating no pain, 10 indicating severe pain, and the middle part indicating varying degrees of pain.
To evaluate the efficacy of Botulinum Toxin Type A for Injection (HengLi®) following multiple doses. | from date of randomization until the date of no response(improvement in VAS score from baseline < 50% )or date of study completion,whichever came first,assessed up to 52 weeks
  Change in mean visual analogue scale (VAS) score of one week from the mean VAS score over one-week at baseline in subjects under continued observation for duration of response to a single dose in the extension period, every 4 week from Week 16 (i.e., Week 16, 20, 24, and so on) until no response (improvement in VAS score from baseline < 50%) or completion of the study.for VAS,Pain was scored on a scale of 0 to10, with 0 indicating no pain, 10 indicating severe pain, and the middle part indicating varying degrees of pain.
To evaluate the efficacy of Botulinum Toxin Type A for Injection (HengLi®) following multiple doses. | from date of randomization until the date of next dose or date of study completion,whichever came first,assessed up to 52 weeks
  Change in visual analogue scale (VAS) score of one week from the mean VAS score over one-week at baseline in subjects receiving additional doses in the extension period, every 4 week after each dose (i.e., 4 week, 8 week, 12 week, and so on) until the next dose or completion of the study;for VAS,Pain was scored on a scale of 0 to10, with 0 indicating no pain, 10 indicating severe pain, and the middle part indicating varying degrees of pain.
To evaluate the efficacy of Botulinum Toxin Type A for Injection (HengLi®) following multiple doses. | from date of randomization until the date of no response(improvement in VAS score from baseline < 50% )or date of study completion,whichever came first,assessed up to 52 weeks
  Change in mean number of daily pain episodes of one week from the mean number of daily pain episodes over one week at baseline in subjects under continued observation for duration of response to a single dose in the extension period, every 4 weeks from Week 16 (i.e., Week 16, 20, 24, and so on) until no response (improvement in visual analogue scale (VAS) score from baseline < 50%) or completion of the study;
To evaluate the efficacy of Botulinum Toxin Type A for Injection (HengLi®) following multiple doses. | from date of randomization until the date of next dose or date of study completion,whichever came first,assessed up to 52 weeks
  Change in mean number of daily pain episodes of one week from the mean number of daily pain episodes over one week at baseline in subjects receiving additional doses in the extension period, every 4 week after each dose (i.e., 4 week, 8 week, 12 week, and so on) until the next dose or completion of the study;
To evaluate the efficacy of Botulinum Toxin Type A for Injection (HengLi®) following multiple doses. | from date of randomization until the date of no response(improvement in VAS score from baseline < 50% )or date of study completion,whichever came first,assessed up to 52 weeks
  Change in mean daily pain duration of subjects with persistent pain over one week [only those with persistent pain (such as dull pain) judged by investigator] from the mean daily pain duration over one week at baseline among subjects under continued observation for duration of response to a single dose in the extension period, every 4 week from Week 16 (i.e., Week 16, 20, 24, and so on) until no response (improvement in visual analogue scale (VAS)score from baseline < 50%) or completion of the study;

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China